CLINICAL TRIAL: NCT05153174
Title: Safety, Feasibility and Efficacy of Sulforaphane (Avmacol) in Chronic Kidney Disease
Brief Title: Study of Sulphoraphane in Chronic Kidney Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Thu Le, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00006759; 1R01DK128677-01 (NIH)
Record Dates: First submitted 2021-11-29; First posted 2021-12-10 (Actual); Results first posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Chronic Kidney Disease stage3; Chronic Kidney Disease stage4
MeSH Terms: interventions — sulforaphane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 2 tablets of Sulforaphane (Experimental): Participants will be given 2 extra strength tablets per day
  Interventions: Drug: Sulforaphane
- 4 tablets of Sulforaphane (Experimental): Participants will be given 4 extra strength tablets per day
  Interventions: Drug: Sulforaphane

INTERVENTIONS:
Drug: Sulforaphane — This is an over-the counter nutritional supplement. Participants will be given the extra strength tablets.
  Other Names: Avmacol

SUMMARY:
The purpose of this study is to test the safety of the compound sulforaphane that boosts the activity of antioxidant genes in the body to combat oxidative stress. Oxidative stress has been shown experimentally to play a role in kidney disease. This drug has been tested in patients with breast cancer who have normal kidney function, but has never been tested in patients with kidney disease.

In this study, the investigators will establish a safe dose for patients with chronic kidney disease based on blood levels achieved in patients with normal kidney function.

DETAILED DESCRIPTION:
We hypothesize that daily intake of sulforaphane (Avmacol Extra Strength (ES)) can decrease kidney disease progression rate and decrease markers of oxidative stress and inflammation in chronic kidney disease (CKD) patients. To test our hypothesis, we will first perform a randomized, Phase 1 clinical trial in a single center funded by an R01 NIDDK award. This is an interventional pharmacokinetic trial, with subjects randomized to different doses of Avmacol ES.

ELIGIBILITY:
Inclusion Criteria:

* eGFR ≥ 20 and <60 ml/min/m2/year, and a decline in eGFR of ≥ 3 ml/min/m2/year in the previous 12 months
* Blood pressure <140/90 mm Hg prior to initiation of sulphoraphane
* stable anti-hypertensive regimen for at least one month prior to initiation of sulphoraphane or successful run-in period
* able to provide consent
* able to swallow capsules

Exclusion Criteria:

* significant co-morbid conditions with life expectancy of <1 year
* uncontrolled hypertension
* serum potassium of >5.5 mEq/L at screening
* New York Heart Association Class 3 or 4 heart failure symptoms, known EF ≤30% or hospital admission for heart failure within the past 3 months
* factors judged to limit adherence to interventions
* current participation in another study
* pregnancy or planning to become pregnant or currently breastfeeding
* history of dementia
* on anticoagulants or immunosuppression
* under treatment for cancer

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thu H Le, MD, FAHA, Principal Investigator — Division of Nephrology Chief
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared after publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: May 2024 data is available. End date to be determined.
Access Criteria: clinicaltrials.gov

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 patient was withdrawn for screen failure before randomizing to an Arm. eGFR (Estimated Glomerular Filtration Rate) lab value was stable & out of eligibility range. 2 patients were randomized to a 6-tablet Arm which was removed in the final Protocol Amendment due to moderate side effects.
Period: Overall Study
Arm/Group | 2 Tablets of Sulforaphane | 4 Tablets of Sulforaphane
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2 Tablets of Sulforaphane | 4 Tablets of Sulforaphane | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (10.3327359445) | 64 (11.1698447661) | 64.4 (10.256793556417)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 6 | 4 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 9 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 6 | 8 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18
Glutathione S-Transferase Mu 1 (GSTM1) Genotype [Count of Participants; unit: Participants] — Collection by buccal swab. GSTM1(0/0) Null genotype compared to those carrying the active GSTM1 (1/1 or 1/0) allele.
  Participants
    GSTM1 (1/1 or 1/0) Allele | 4 | 4 | 8
    GSTM1 (0/0) Null | 5 | 5 | 10
Stage of Chronic Kidney Disease (CKD) [Count of Participants; unit: Participants] — eGFR=Estimated Glomerular Filtration Rate, based on Creatinine level.
  Participants
    Stage 3 CKD (eGFR 30-59) | 8 | 7 | 15
    Stage 4 CKD (eGFR 15-29) | 1 | 2 | 3
Estimated Glomerular Filtration Rate (eGFR) level at Baseline [Mean (Full Range); unit: mL/min/1.73 m2] | 33.3 [28 to 39] | 34.6 [28 to 44] | 34.2 [28 to 44]

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-Time Curve (AUC 0-8h) in Plasma
Description: Sulforaphane drug levels will be measured in plasma at 0, 1, 2, 4, and 8 hours.
Time Frame: prior to initial dose on day 7 and 1, 2, 4, and 8 hours post-dose
Population: First 6 samples (2 from each arm) not included due to problem with standards resulting in no absolute quantification.
Measure: Mean (Standard Deviation); unit: nmol h/L
Arm/Group | 2 Tablets of Sulforaphane | 4 Tablets of Sulforaphane
Number analyzed (Participants) | 7 | 7
nmol h/L | 700.0 (376.5) | 718.4 (335.8)
Statistical Analysis 1: Comparison: 2 Tablets of Sulforaphane vs 4 Tablets of Sulforaphane; Test type: Equivalence — p < 0.05 to reject null hypothesis of equivalence; p = 0.931, t-test, 2 sided

2. Primary Outcome: Area Under the Concentration-Time Curve (AUC 0-8h) in Urine
Description: Sulforaphane drug levels will be measured in urine at 0, 1, 2, 4, and 8 hours.
Time Frame: prior to initial dose on day 7 and 1, 2, 4, and 8 hours post-dose
Population: First 6 samples (2 from each arm) not included due to problem with standards resulting in no absolute quantification.
Measure: Mean (Standard Deviation); unit: nmol h/L
Arm/Group | 2 Tablets of Sulforaphane | 4 Tablets of Sulforaphane
Number analyzed (Participants) | 7 | 7
nmol h/L | 12497.0 (9569.2) | 24928.8 (23028.8)
Statistical Analysis 1: Comparison: 2 Tablets of Sulforaphane vs 4 Tablets of Sulforaphane; Test type: Equivalence — p < 0.05 to reject null hypothesis of equivalence; p = 0.224, t-test, 2 sided

3. Primary Outcome: Number of Participants With an Adverse Event
Description: Adverse Event is any side effect outside of the subject's baseline.
Time Frame: day 7
Measure: Count of Participants; unit: Participants
Arm/Group | 2 Tablets of Sulforaphane | 4 Tablets of Sulforaphane
Number analyzed (Participants) | 9 | 9
Participants | 5 | 7

ADVERSE EVENTS:
Time Frame: 10 months, 11 days
Description: Health symptoms that differ from the individual's baseline. Anticipated AE's include gastrointestinal symptoms.
Arm/Group | 2 Tablets of Sulforaphane | 4 Tablets of Sulforaphane
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 4/9 | 7/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 2 Tablets of Sulforaphane (N=9) | 4 Tablets of Sulforaphane (N=9)
Nausea (Gastrointestinal disorders) | 0 | 4
Diarrhea, or Loose Stool (Gastrointestinal disorders) | 2 | 2
Flatus (Gas) (Gastrointestinal disorders) | 1 | 3
Bloated Stomach (Gastrointestinal disorders) | 0 | 3
Heartburn/Reflux (Gastrointestinal disorders) | 0 | 2
Indigestion/Abdominal Pain (Gastrointestinal disorders) | 1 | 3

LIMITATIONS AND CAVEATS:
At the time of review with the Data Safety Monitoring Committee, the study had consented 21 patients and enrolled 18 patients out of 24 targeted. 2 of the 21 patients were randomized to a 6-tablet Arm, which was removed in the final Protocol Amendment due to moderate side effects/adverse events. 1 patient withdrew before study procedures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-17): https://cdn.clinicaltrials.gov/large-docs/74/NCT05153174/Prot_SAP_000.pdf
  • Informed Consent Form (2022-12-09): https://cdn.clinicaltrials.gov/large-docs/74/NCT05153174/ICF_001.pdf